CLINICAL TRIAL: NCT02108301
Title: Hepatitis C in Renal Transplant Recipients - Safety and Efficacy of a Conversion of Immunosuppression to High-dose Cyclosporine A and Its Impact on Hepatitis C Virus-replication, Parameters of Liver Function and Glucose Tolerance. An Open Label Trial.
Brief Title: Hepatitis C in Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. Alice Schmidt (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Alice Schmidt, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK477/2011
Record Dates: First submitted 2014-04-01; First posted 2014-04-09 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Hepatitis C-virus Infection; Renal Transplantation
Keywords: chronic hepatitis C-virus infection; renal transplantation; glucose tolerance; immunosuppression

ARMS (1):
- tacrolimus-cyclosporine A (Experimental): conversion of immunosuppression from tacrolimus to cyclosporine A in hepatitis C-positive renal transplant recipients
  Interventions: Drug: tacrolimus-cyclosporine A

INTERVENTIONS:
Drug: tacrolimus-cyclosporine A — conversion of immunosuppression from tacrolimus to cyclosporine A in hepatitis C-positive renal transplant recipients

SUMMARY:
The aim of the present trial is to evaluate whether the conversion of immunosuppression from tacrolimus to cyclosporine A induces changes in (i) hepatitis C-virus load, (ii) parameters of hepatic function and (iii) parameters of glucose tolerance in hepatitis C-positive renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* prior renal transplantation
* current tacrolimus-based immunosuppressive regimen
* hepatitis C-infection
* age 18-70 years

Exclusion Criteria:

* current hemodialysis or peritoneal dialysis
* pregnancy or breastfeeding
* known contraindication for cyclosporine A-treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change in Hepatitis C-virus load at 12 weeks | one day before and 4, 8 and 12 weeks after the conversion

SECONDARY OUTCOMES:
change in oral glucose insulin sensitivity (OGIS) index at 12 weeks | one day before and 12 weeks after the conversion
change in serum hepcidin levels at 12 weeks | one day before and 12 weeks after the conversion

OTHER OUTCOMES:
serum creatinine levels | 12 weeks
serum glutamic-pyruvic transaminase concentrations | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Handisurya A, Kerscher C, Tura A, Herkner H, Payer BA, Mandorfer M, Werzowa J, Winnicki W, Reiberger T, Kautzky-Willer A, Pacini G, Saemann M, Schmidt A. Conversion from Tacrolimus to Cyclosporine A Improves Glucose Tolerance in HCV-Positive Renal Transplant Recipients. PLoS One. 2016 Jan 6;11(1):e0145319. doi: 10.1371/journal.pone.0145319. eCollection 2016. PMID 26735686